CLINICAL TRIAL: NCT02718560
Title: Effectiveness of Intensive Handwriting Rehabilitation in Subjects With Parkinson's Disease
Brief Title: Handwriting Rehabilitation in Parkinson Disease
Acronym: HRPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Handwriting rehab in PD
Record Dates: First submitted 2016-03-15; First posted 2016-03-24 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Parkinson Disease; Neurorehabilitation; Handwriting
MeSH Terms: conditions — Parkinson Disease | interventions — Functional Laterality

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 - Writing with 1 cm cue (Experimental): This group uses to write space of 1 cm size
  Interventions: Behavioral: Writing
- Group 2 - Writing with 1.5 cm cue (Experimental): This group uses to write space of 1.5 cm size
  Interventions: Behavioral: Writing
- Group 3 - Writing without cue (Experimental): This group writes without using cues
  Interventions: Behavioral: Writing
- Group 4 - no writing (No Intervention): This group do not write. Only wrist mobilization is performed.

INTERVENTIONS:
Behavioral: Writing — Writing exercise with or without cues for 1 hour per day for 4 days at week for 4 weeks
  Arms: Group 1 - Writing with 1 cm cue; Group 2 - Writing with 1.5 cm cue; Group 3 - Writing without cue

SUMMARY:
The aim of the study is to evaluate the efficacy of an intensive handwriting treatment in Parkinson's Disease.

DETAILED DESCRIPTION:
The investigators aimed to understand whether an intensive handwriting treatment with cognitive engagement is more effective than a treatment exploiting only the passive wrist joint mobilization in Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease patients

Exclusion Criteria:

* Mini Mental State Examination (MMSE) score < 24
* Left handed subjects
* Subjects with dyskinesias
* Subjects with Deep Brain Stimulation

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
letters size | 4 weeks

SECONDARY OUTCOMES:
writing speed (time spent to write every single letter and word, measured in milliseconds) | 4 weeks
centimeters away from a straight line during writing | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Ospedale Generale Di Zona Moriggia-Pelascini
Locations (1):
- Ospedale Generale di zona Moriggia Pelascini, Gravedona Ed Uniti, Como, Italy

IPD SHARING:
Plan to Share IPD: No